CLINICAL TRIAL: NCT07046676
Title: Research on the Application of Sodium Valproate Personalized Medication Based on Pharmacogenetics
Brief Title: Pharmacogenetics-Based Study on Individualized Use of Sodium Valproate
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: nhfy20250317
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Valproic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sodium valproate (Experimental): According to the dosage forms of sodium valproate, they are divided into the sodium valproate tablet group, the sodium valproate oral solution group and the sodium valproate sustained-release tablet group.
  Interventions: Drug: sodium valproate

INTERVENTIONS:
Drug: sodium valproate — All three groups are administered twice a day via oral administration. Patients are given different doses based on their body weight and the therapeutic effect in controlling epilepsy.

SUMMARY:
Sodium valproate (VPA) is a first-line prescription drug widely used in the treatment of epilepsy. However, in clinical applications, it has been found that there is a large individual variation in the blood concentration of VPA. In particular, excessively high blood drug concentrations can lead to various side effects, especially hepatotoxicity. Blood drug concentration monitoring can reduce the toxic and side effects of VPA to a certain extent and improve its effectiveness, but it is too cumbersome. A large number of studies have shown that the efficacy and toxic side effects of VPA are closely related to its in vivo metabolism process. The in vivo metabolism of VPA is affected by many factors, and the genetic polymorphism of drug-metabolizing enzymes is an important factor leading to differences in blood drug concentrations and affecting the dosage of VPA. The three products generated by the biotransformation of VPA by CYP450 enzymes are all related to hepatotoxicity. The formation of 4-ene-VPA is largely catalyzed by CYP2C9 and CYP2A6. Mutations in the CYP2A6 gene may be related to VPA hepatotoxicity, but there is a lack of further direct evidence. 50% of VPA in the body is acidified and metabolized into inactive products by uridine diphosphate glucuronosyltransferase (UGT) through phase II conjugation reactions. However, there is evidence that the genetic polymorphism of UGT can significantly affect the blood drug concentration of metformin. Based on the above research, we selected CYP2A6, UGT1A6, etc. as candidate genes, and studied the impact of genetic polymorphisms on the individual differences of sodium valproate through association analysis, with the hope of establishing a genetic model for optimal dosage and providing new strategies for the individualized use of VPA.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with epilepsy (primary epilepsy, secondary epilepsy) and with complete clinical data
* Regular use of valproic acid sodium for at least 5 days (with blood drug concentration reaching a steady state) and strong medication compliance
* Patients using combined anti-epileptic drugs or using valproic acid sodium alone
* Patients without significant liver or kidney dysfunction, and not in the pregnancy period

Exclusion Criteria:

* Patients with incomplete data, poor compliance, and those whose blood drug concentration was not measured at the correct concentration
* Patients with major respiratory, gastrointestinal, liver, kidney or other serious diseases
* Patients using valproic acid solely for epilepsy prevention
* Patients who have used valproic acid for more than 5 days but have frequently changed the dosage form during the process
* Patients over 65 years old and in the 1CU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
The blood concentration of valproic acid | Collect data on the first patient and follow up for a period of three years.
  The effective blood concentration of valproic acid should be maintained at 50 - 100 ug/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of South China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: No